CLINICAL TRIAL: NCT00130728
Title: A Phase III, Multicenter, Placebo-Controlled, Double-Blind, Randomized Clinical Trial to Evaluate the Efficacy of Bevacizumab in Combination With Tarceva (Erlotinib) Compared With Tarceva Alone for Treatment of Advanced Non-Small Cell Lung Cancer (NSCLC) After Failure of Standard First-Line Chemotherapy
Brief Title: A Study to Evaluate the Efficacy of Bevacizumab in Combination With Tarceva for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSI3364g
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Avastin; Tarceva; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- erlotinib HCl + bevacizumab (Experimental): oral erlotinib HCl 150 mg/day orally + intravenous infusion of bevacizumab at a dose of 15 mg/kg on the first day of each 3-week cycle
  Interventions: Drug: bevacizumab
- erlotinib HCl + placebo (Placebo Comparator): oral erlotinib HCl 150 mg/day orally + intravenous infusion of placebo at a dose of 15 mg/kg on the first day of each 3-week cycle
  Interventions: Drug: erlotinib HCl; Drug: placebo

INTERVENTIONS:
Drug: bevacizumab — intravenous infusion of bevacizumab at a dose of 15 mg/kg on the first day of each 3-week cycle
  Arms: erlotinib HCl + bevacizumab
Drug: erlotinib HCl — oral erlotinib HCl 150 mg/day orally
  Arms: erlotinib HCl + placebo
Drug: placebo — intravenous infusion of placebo at a dose of 15 mg/kg on the first day of each 3-week cycle
  Arms: erlotinib HCl + placebo

SUMMARY:
This is a Phase III, multicenter, placebo-controlled, double-blind, randomized study. Approximately 650 patients will be randomized in a 1:1 ratio to one of two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Cytologically or histologically confirmed NSCLC
* Clinical or radiographic progression during or after first-line chemotherapy or chemoradiotherapy for NSCLC
* Consent to provide archival tissue for analysis is required for participation in this study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Age ≥ 18 years
* Use of an acceptable means of contraception for men and women of childbearing potential
* International normalized ratio (INR) no greater than 1.3 and an aPTT no greater than the upper limits of normal within 28 days prior to enrollment for patients not on low-molecular-weight heparin or fondaparinux

Exclusion Criteria:

* Squamous cell carcinoma
* Prior treatment with an investigational or marketed inhibitor of the Epidermal Growth Factor Receptor (EGFR) pathway or anti-angiogenesis agent
* Systemic chemotherapy, radiotherapy, or investigational treatment within 28 days prior to randomization
* Local palliative radiotherapy within 14 days prior to randomization or persistent adverse effects from radiotherapy that have not resolved to Grade 2 or less following completion of treatment
* Whole brain radiotherapy or stereotactic radiosurgery for brain metastases within 4 weeks of Day 0
* Neurosurgery for brain metastases within 24 weeks of Day 0
* Brain biopsy within 12 weeks of Day 0
* Current use of dexamethasone for treatment associated with brain metastases
* History of gross hemoptysis within 3 months prior to randomization unless definitively treated with surgery or radiation
* History of any of the following within 6 months prior to Day 0: serious systemic disease, uncontrolled hypertension, unstable angina, New York Heart Association (NYHA) Grade 2 or greater Congestive Heart Failure (CHF), unstable symptomatic arrhythmia requiring medication, clinically significant peripheral vascular disease, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Evidence of bleeding diathesis or coagulopathy or other serious or acute internal bleeding within 6 months prior to randomization
* Central Nervous System (CNS) bleeding; history or clinical evidence of CNS stroke (hemorrhagic or thrombotic) within the last 6 months
* Progressive neurologic symptoms in patients with a history of brain metastases
* Full-dose anticoagulation with warfarin
* Chronic daily use of aspirin or other full-dose nonsteroidal anti-inflammatory drugs (NSAIDs) with anti-platelet activity
* In-patient surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
* Minor surgical procedure, fine needle aspirations or core biopsy within 7 days prior to randomization
* Anticipation of need for a major surgical procedure during the course of the study
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to take oral medication or requirement for intravenous (IV) alimentation or total parenteral nutrition with lipids, or prior surgical procedures affecting absorption
* Pregnancy or breast-feeding
* Presence of another invasive cancer within 5 years prior to randomization
* Evidence of confusion or disorientation, or history of major psychiatric illness that may impair the patient's understanding of the Informed Consent Form or their ability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2005-06-08 (Actual); Primary Completion 2008-07-15 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Kaiser Permanente - Vallejo, Vallejo, California
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Anne Arundel Health System Research Instit-Annapolis Oncology Ctr, Annapolis, Maryland

REFERENCES:
- [Derived] Herbst RS, Ansari R, Bustin F, Flynn P, Hart L, Otterson GA, Vlahovic G, Soh CH, O'Connor P, Hainsworth J. Efficacy of bevacizumab plus erlotinib versus erlotinib alone in advanced non-small-cell lung cancer after failure of standard first-line chemotherapy (BeTa): a double-blind, placebo-controlled, phase 3 trial. Lancet. 2011 May 28;377(9780):1846-54. doi: 10.1016/S0140-6736(11)60545-X. PMID 21621716

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
Started | 319 | 317
Received Study Drug (Safety Population) | 313 | 313
Completed | 57 | 57
Not Completed | 262 | 260
Not completed — Death | 258 | 258
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo | Total
Number analyzed (Participants) | 319 | 317 | 636
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.4) | 65.0 (10.3) | 64.9 (10.4)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 59 years | 91 | 90 | 181
  Between 60 and 64 years | 62 | 66 | 128
  Between 65 and 69 years | 59 | 53 | 112
  >= 70 years | 107 | 108 | 215
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 147 | 295
  Male | 171 | 170 | 341

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Among All Randomized Patients
Description: Overall Survival was defined as the period from the date of randomization until the date of patient death from any cause. For patients who had not died, survival data was censored at the date of last contact.
Time Frame: From the date of randomization until the date of patient death from any cause, or the date of last contact. (Up to 3.1 years)
Population: Randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
Number analyzed (Participants) | 319 | 317
months | 9.3 [7.39 to 11.47] | 9.2 [7.85 to 11.60]
Statistical Analysis 1: Comparison: Erlotinib HCl + Bevacizumab vs Erlotinib HCl + Placebo; Test type: Superiority or Other; p = 0.7583, Log Rank — relative to placebo arm; Hazard Ratio (HR) = .970, 95% CI [0.799 to 1.177] — Stratified analysis; Hazard ratio is relative to placebo arm

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to documented disease progression, as determined by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST), or death on study treatment, whichever occurred first.
Time Frame: From randomization to documented disease progression or death on study treatment, whichever occurred first. (Up to 3.1 years)
Population: Randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
Number analyzed (Participants) | 319 | 317
months | 3.4 [2.79 to 4.27] | 1.7 [1.48 to 2.53]
Statistical Analysis 1: Comparison: Erlotinib HCl + Bevacizumab vs Erlotinib HCl + Placebo; Test type: Superiority or Other; p < .0001, Log Rank — relative to placebo arm; Hazard Ratio (HR) = 0.623, 95% CI [0.519 to 0.748] — Stratified analysis; hazard ratio is relative to placebo arm

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as a complete or partial response determined by RECIST on two consecutive occasions >= 4 weeks apart.
Time Frame: The median duration of Objective response was up to 9.7 months
Population: Only patients with measurable disease at baseline were included in the analysis of the objective response. Patients without a post-baseline tumor assessment were considered non-responder.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
Number analyzed (Participants) | 301 | 306
Percentage of participants | 12.6 [9.1 to 16.8] | 6.2 [3.8 to 9.5]
Statistical Analysis 1: Comparison: Erlotinib HCl + Bevacizumab vs Erlotinib HCl + Placebo; Test type: Superiority or Other; p = 0.0068, Mantel Haenszel — Relative to placebo arm; Percentage difference = 6.4, 95% CI [1.8 to 11.3] — Difference in objective response rates relative to placebo arm

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the period from the date of the initial partial or complete response until the date of disease progression or death on study treatment from any cause. For patients who had not died, data was censored at the date of last contact.
Time Frame: Period from Objective response until disease progression or death on study treatment. (Up to 29.5 months)
Population: Patients with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
Number analyzed (Participants) | 38 | 19
months | 9.7 [6.90 to 19.48] | 8.4 [3.48 to 14.88]

ADVERSE EVENTS:
Time Frame: From randomization to up to 3.8 years (for Adverse Events) From randomization until last patient last visit or up to 14.5 years from start of study (for Serious Adverse Events)
Description: Safety Evaluable Population
Arm/Group | Erlotinib HCl + Bevacizumab | Erlotinib HCl + Placebo
All-Cause Mortality (participants affected / at risk) | 258/313 | 258/313
Serious Adverse Events (participants affected / at risk) | 146/313 | 121/313
Other Adverse Events (participants affected / at risk) | 310/313 | 306/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib HCl + Bevacizumab (N=313) | Erlotinib HCl + Placebo (N=313)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Acute Myocardial Infarction (Cardiac disorders) | 4 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 4
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 5 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Blindness Unilateral (Eye disorders) | 1 | 0
Retinal Haemorrhage (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastritis Erosive (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrointestinal Perforation (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal Perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 2 | 1
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 3 | 2
Death (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 4
Pyrexia (General disorders) | 3 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Food Allergy (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Breast Cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 2 | 3
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Empyema (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 2 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 1 | 0
Perirectal Abscess (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 15 | 10
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 3
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation Retinopathy (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tracheal Injury (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Blood Culture Positive (Investigations) | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 1
Liver Function Test Abnormal (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 3
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 3 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Intracranial Pressure Increased (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 2 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Toxic Encephalopathy (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 2
Mental Status Changes (Psychiatric disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 24
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 6
Hypertension (Vascular disorders) | 4 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Jugular Vein Thrombosis (Vascular disorders) | 1 | 1
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Trousseau's Syndrome (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea Infectious (Gastrointestinal disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib HCl + Bevacizumab (N=313) | Erlotinib HCl + Placebo (N=313)
Anaemia (Blood and lymphatic system disorders) | 19 | 29
Diarrhoea (Gastrointestinal disorders) | 203 | 162
Nausea (Gastrointestinal disorders) | 121 | 99
Vomiting (Gastrointestinal disorders) | 57 | 49
Constipation (Gastrointestinal disorders) | 49 | 45
Stomatitis (Gastrointestinal disorders) | 40 | 27
Abdominal Pain (Gastrointestinal disorders) | 29 | 25
Dyspepsia (Gastrointestinal disorders) | 21 | 16
Dysphagia (Gastrointestinal disorders) | 19 | 12
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 18 | 10
Fatigue (General disorders) | 146 | 124
Pyrexia (General disorders) | 33 | 23
Asthenia (General disorders) | 34 | 20
Chest Pain (General disorders) | 27 | 24
Oedema Peripheral (General disorders) | 18 | 32
Mucosal Inflammation (General disorders) | 35 | 16
Pain (General disorders) | 15 | 18
Chills (General disorders) | 23 | 11
Urinary Tract Infection (Infections and infestations) | 33 | 26
Upper Respiratory Tract Infection (Infections and infestations) | 30 | 30
Pneumonia (Infections and infestations) | 9 | 16
Bronchitis (Infections and infestations) | 10 | 18
Sinusitis (Infections and infestations) | 16 | 8
Weight Decreased (Investigations) | 65 | 41
Anorexia (Metabolism and nutrition disorders) | 104 | 75
Dehydration (Metabolism and nutrition disorders) | 35 | 24
Decreased Appetite (Metabolism and nutrition disorders) | 36 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 46 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 27
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 34 | 23
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 24 | 20
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 19 | 15
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 16 | 17
Headache (Nervous system disorders) | 53 | 28
Dizziness (Nervous system disorders) | 41 | 31
Dysgeusia (Nervous system disorders) | 29 | 19
Insomnia (Psychiatric disorders) | 38 | 25
Anxiety (Psychiatric disorders) | 26 | 30
Depression (Psychiatric disorders) | 31 | 19
Proteinuria (Renal and urinary disorders) | 18 | 8
Dysuria (Renal and urinary disorders) | 16 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 76
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 61 | 64
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 63 | 30
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 27 | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 33 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 22 | 14
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Rash (Skin and subcutaneous tissue disorders) | 193 | 184
Dry Skin (Skin and subcutaneous tissue disorders) | 63 | 58
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 58 | 42
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 40
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 16
Erythema (Skin and subcutaneous tissue disorders) | 16 | 11
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 8 | 16
Hypertension (Vascular disorders) | 77 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study.

DOCUMENTS (2):
  • Study Protocol (2012-10-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT00130728/Prot_000.pdf
  • Statistical Analysis Plan (2006-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT00130728/SAP_001.pdf